CLINICAL TRIAL: NCT04850963
Title: Effects of Dualsite Anodic tDCS on Lower Limbs Function in Patients After Stroke
Brief Title: Effects of Dualsite Anodic tDCS on Lower Limbs Function in Patients After Stroke: Randomized, Double-blind, Placebo-controlled, Crossover Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AVCtDCS
Record Dates: First submitted 2021-03-24; First posted 2021-04-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Chronic
Keywords: Stroke; Transcranial direct current stimulation
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - anodal tDCS (Active Comparator): Participants will receive 10 tDCS sessions, for 20 minutes, on days alternate (3 times a week).
  The neurostimulator TCT-Research will be used for stimulation. The electrodes will be positioned according to the international classification system of the electroencephalogram 10/20. For group 1 (anodic tDCS) the anodic electrode (5x5 cm) will be applied to the primary motor area (C3/C4) ipsilateral to the lesion and the reference electrode (6x9 cm) to the deltoid muscle region.
  Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  Interventions: Device: Transcranial direct current stimulation (tDCS dualsite) + dual-task traning; Device: Transcranial direct current stimulation sham + dual-task training
- Group 2 - tDCS dualsite (Active Comparator): Participants will receive 10 tDCS sessions, for 20 minutes, on days alternate (3 times a week).
  The neurostimulator TCT-Research will be used for stimulation. The electrodes will be positioned according to the international classification system of the electroencephalogram 10/20. In group 2 (dualsite tDCS) two active electrodes (5x5 cm) will be used, which will be positioned over the primary motor area (C3/C4) and over the dorsolateral prefrontal cortex (F3 or F4) in the ipsilateral hemisphere. For this stimulation modality, two active electrodes (anodic) and a reference electrode (6x9 cm) will be used on the deltoid muscle region.
  Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  Interventions: Device: Transcranial direct current stimulation (Anodal tDCS) + dual-task training; Device: Transcranial direct current stimulation sham + dual-task training
- Group 3 - tDCS sham (Placebo Comparator): Participants will receive 10 tDCS sessions, for 20 minutes, on days alternate (3 times a week).
  The neurostimulator TCT-Research will be used for stimulation. The electrodes will be positioned according to the international classification system of the electroencephalogram 10/20. For group 3 (simulated tDCS) the positioning of the electrodes will be the same as for group 1, however the device will be configured in sham mode in which the current will cease 30 seconds after the start of stimulation.
  Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  Interventions: Device: Transcranial direct current stimulation (Anodal tDCS) + dual-task training; Device: Transcranial direct current stimulation (tDCS dualsite) + dual-task traning

INTERVENTIONS:
Device: Transcranial direct current stimulation (Anodal tDCS) + dual-task training — anodal tDCS 837 / 5.000 Resultados de tradução Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training, which will include: (1) walking repeating phrases spoken by the researcher; (2) walking counting numbers in ascending order; (3) walk while counting the numbers in descending order; (4) walking during the execution of a string of words; (5) Walking while listening to a list of fruits and saying "YES" when hearing the word "strawberry" and (6) walking reciting a phrase backwards. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  The tasks will be performed performing forward, side and back march. Subjects will be instructed to focus on both tasks. The training will have a total duration of 20 minutes in each session.
  Other Names: anodal tDCS
  Arms: Group 2 - tDCS dualsite; Group 3 - tDCS sham
Device: Transcranial direct current stimulation (tDCS dualsite) + dual-task traning — tDCS dualsite 837 / 5.000 Resultados de tradução Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training, which will include: (1) walking repeating phrases spoken by the researcher; (2) walking counting numbers in ascending order; (3) walk while counting the numbers in descending order; (4) walking during the execution of a string of words; (5) Walking while listening to a list of fruits and saying "YES" when hearing the word "strawberry" and (6) walking reciting a phrase backwards. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  The tasks will be performed performing forward, side and back march. Subjects will be instructed to focus on both tasks. The training will have a total duration of 20 minutes in each session.
  Other Names: tDCS dualsite
  Arms: Group 1 - anodal tDCS; Group 3 - tDCS sham
Device: Transcranial direct current stimulation sham + dual-task training — tDCS sham 837 / 5.000 Resultados de tradução Simultaneously with the tDCS sessions, participants will be submitted to a physical therapy protocol based on motor and cognitive dual-task training, which will include: (1) walking repeating phrases spoken by the researcher; (2) walking counting numbers in ascending order; (3) walk while counting the numbers in descending order; (4) walking during the execution of a string of words; (5) Walking while listening to a list of fruits and saying "YES" when hearing the word "strawberry" and (6) walking reciting a phrase backwards. Each task will have a duration of 3 minutes, followed by a rest period of 30s.
  The tasks will be performed performing forward, side and back march. Subjects will be instructed to focus on both tasks. The training will have a total duration of 20 minutes in each session.
  Other Names: tDCS sham
  Arms: Group 1 - anodal tDCS; Group 2 - tDCS dualsite

SUMMARY:
It is currently known that Transcranial Direct Current Stimulation (tDCS) can modulate cortical activity, being considered an important resource in the treatment of sequelae resulting from stroke. However, evidence of the effects of tDCS on lower limb motor recovery after stroke remains scarce and inconclusive. Furthermore, little is known about the effects of dualsite tDCS in chronic patients. Therefore, the present study seeks to compare the effects of conventional anodic tDCS (M1) with double-site/dualsite anodic tDCS (M1 + DLPFC) and simulated tDCS on lower limb motor function in patients after ischemic stroke in a chronic stage. The study is a randomized, double-blind, placebo-controlled, crossover clinical trial with subjects after stroke. After recruitment and initial screening, participants will be randomized into three groups: G1: anodic tDCS - participants who will receive real current over the primary motor area; G2: dualsite tDCS - participants who will receive real current over the primary motor area and dorsolateral prefrontal area (DLPFC) and G3: simulated tDCS - participants who will receive simulated stimulation. Participants will receive 10 tDCS sessions, for 20 minutes, associated with a physical therapy protocol based on a dual motor and cognitive task, on alternate days (3 times a week). In each phase of the study, pre- and post-intervention evaluations will be carried out, the evaluated outcomes will be: motor function (Fugl-Meyer Scale), functional connectivity (EEG), quality of life (EQ-5D), level of functional disability ( Rankin Scale), static balance (Biodex Balance System) and cognitive function (MoCA). Statistical analyzes will be performed using SPSS software (Version 20.0) and MATLAB 9.2.0 with a significance level of p <0.05.

DETAILED DESCRIPTION:
Participants will be divided into 03 groups: G1: anodic tDCS - participants who will receive real current over the primary motor area; G2: dualsite tDCS - participants who will receive real current over the primary motor area and over the dorsolateral prefrontal area (DLPFC) and G3: simulated tDCS - participants who will receive simulated stimulation. Participants will be entered into the study through the eligibility criteria and will be randomly allocated, with block exchange at a rate of 1:1:1.

In each phase of the study, participants will receive 10 tDCS sessions, for 20 minutes, on alternate days (3 times a week, excluding weekends). The TCT-Research neurostimulator will be used for stimulation. The electrodes will be positioned according to the 10-20 international electroencephalogram classification system. Electrodes wrapped in sponges, moistened with saline solution (0.9% NaCl) will be used. The applied current will be 2mA (5x5 cm active electrodes; 25 cm2; current density of 0.08 mA/cm2).

For group 1 (anodic tDCS) the anodic electrode (5x5 cm) will be applied to the primary motor area (C3/C4) ipsilateral to the lesion and the reference electrode (6x9 cm) to the deltoid muscle region. In group 2 (dualsite tDCS) two active electrodes (5x5 cm) will be used, which will be positioned over the primary motor area (C3/C4) and over the dorsolateral prefrontal cortex (F3 or F4) in the ipsilateral hemisphere. For this stimulation modality, two active electrodes (anodic) and a reference electrode (6x9 cm) will be used on the deltoid muscle region.

For group 3 (simulated tDCS) the positioning of the electrodes will be the same as for group 1, however the device will be configured in sham mode in which the current will cease 30 seconds after the start of stimulation, in this way the effects of active stimulation will be simulated and the participants will perceive the sensations typically felt, but without the induction of clinical effects (Nitsche & Paulus, 2000). At the end of each session, participants will be asked to report any unpleasant effects and asked about possible adverse effects. In addition, all participants will be blind to the type of stimulation they will receive.

ELIGIBILITY:
Inclusion Criteria:

* Single episode of unilateral, ischemic stroke in middle cerebral artery proven by means of magnetic resonance imaging or computed tomography.
* Classification of brain injury based on the criteria: Oxfordshire Community Stroke Project (OCSP) or Trial of Org 10172 in Acute Stroke Treatment (TOAST);
* Patients in the chronic stage (after six months after the injury)
* Individuals over 18 years of age;
* Both sexes;
* Absence of mental disorders, assessed using the Self Reporting Questionnaire (SRQ-20), with a cut-off point of 7/8 points.
* Absence of cognitive deficits, assessed using the Mini Mental State Examination (MMSE> 24).
* Patients with mild to moderate degree of injury severity (NIHHS <17 points).

Exclusion Criteria:

* Patients with other associated pathologies that can influence motor activity (example: traumatic brain injury, brain tumor);

  •- Participants unable to complete the initial assessment due to severe aphasia (Token Test <17);
* habitual use of drugs or alcohol;
* Use of drugs that modulate the activity of the Central Nervous System;
* Gestation;
* Use of metallic / electronic implants and / or cardiac pacemakers;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-24 (Estimated); Study Completion 2022-12-24 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer assessment (FMA) pre-intervention (T0) | The evaluations will be carried out in pre-intervention (T0)
  Fugl-Meyer assessment (FMA) for lower limbs pre-intervention (T0)
Fugl-Meyer assessment (FMA) after the stimulation protocol (T1) | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  Fugl-Meyer assessment (FMA) for lower limbs after the stimulation protocol (T1)

SECONDARY OUTCOMES:
Functional connectivity (EEG) pre-intervention (T0) | The evaluations will be carried out in pre-intervention (T0)
  The functional connectivity of the target network will be assessed, through the acquisition of the EEG
Functional connectivity (EEG) after the stimulation protocol (T1) | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  The functional connectivity of the target network will be assessed, through the acquisition of the EEG
EQ-5D (T0) | The evaluations will be carried out in pre-intervention (T0).
  Quality of life. Presenting a final score from 0 to 100, where 0 corresponds to the worst general state of health and 100 the best state of health.
EQ-5D (T1) | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  Quality of life.Presenting a final score from 0 to 100, where 0 corresponds to the worst general state of health and 100 the best state of health.
Modified Rankin Scale pre-intervention (T0) | The evaluations will be carried out in pre-intervention (T0).
  Functional disability. The score on the Rankin scale ranges from 0 to 6, in order to assess the patient's neurological condition, in which the higher the value, the worse the condition.
  0 - No symptoms
  1. - No significant disabilities
  2. - Mild disability
  3. - Moderate disability
  4. - Moderate-severe disability
  5. - Severe disability
  6. - Death
Modified Rankin Scale after the stimulation protocol (T1) | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  Functional disability. The score on the Rankin scale ranges from 0 to 6, in order to assess the patient's neurological condition, in which the higher the value, the worse the condition.
  0 - No symptoms
  1. - No significant disabilities
  2. - Mild disability
  3. - Moderate disability
  4. - Moderate-severe disability
  5. - Severe disability
  6. - Death
Balance | The T0 assessment will be performed up to one week after the stimulation protocol is completed.
  Biodex Balance System (BBS)
Balance | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  Biodex Balance System (BBS)
MoCA | The T0 assessment will be performed up to one week after the stimulation protocol is completed.
  Cognitive function
MoCA | The T1 assessment will be performed up to one week after the stimulation protocol is completed.
  Cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraíba
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No